CLINICAL TRIAL: NCT06923085
Title: Bilateral Sensorimotor Dysfunction in the Upper Extremities in Unilateral Cervical Radiculopathies: A Level-Specific Approach
Brief Title: Upper Extremity Dysfunction in Patients With Cervical Radiculopathy
Acronym: CerRad-UE
Status: Completed | Type: Observational
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Tuba Eren, Lecturer, University of Beykent
Other Study IDs: GO 21/906
Record Dates: First submitted 2025-03-11; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: C4-5 Radiculopathy Group: Patients with confirmed C4-5 cervical radiculopathy. Assessments included pain (VAS), neck disability (NDI), upper extremity functionality (DASH), muscle strength measurements, sensory function, hand performance, kinesiophobia (TAMPA) and emotional status (Beck Inventory).
  Interventions: Other: Observational Assessment Only
- Group 2: C5-6 Radiculopathy Group: Patients with confirmed C5-6 cervical radiculopathy. Assessments included pain (VAS), neck disability (NDI), upper extremity functionality (DASH), muscle strength measurements, sensory function, hand performance, kinesiophobia (TAMPA) and emotional status (Beck Inventory).
  Interventions: Other: Observational Assessment Only
- Group 3: C6-7 Radiculopathy Group: Patients with confirmed C6-7 cervical radiculopathy. Assessments included pain (VAS), neck disability (NDI), upper extremity functionality (DASH), muscle strength measurements, sensory function, hand performance, kinesiophobia (TAMPA) and emotional status (Beck Inventory).
  Interventions: Other: Observational Assessment Only
- Control Group: Control subjects with non-specific neck pain without radiculopathy. Assessments included pain (VAS), neck disability (NDI), upper extremity functionality (DASH), muscle strength measurements, sensory function, hand performance, kinesiophobia (TAMPA) and emotional status (Beck Inventory).
  Interventions: Other: Observational Assessment Only

INTERVENTIONS:
Other: Observational Assessment Only — This is an observational study examining bilateral sensorimotor function in patients with cervical radiculopathy. No interventional procedures were applied. Participants underwent comprehensive assessments including pain evaluation (VAS), neck disability (NDI), upper extremity functionality (DASH), muscle strength measurements, sensory function testing, hand performance evaluation, kinesiophobia (TAMPA), and emotional status assessment (Beck Inventory). The study compared findings between different cervical radiculopathy groups and a control group with non-specific neck pain.

SUMMARY:
This study will examine how cervical radiculopathy (a pinched nerve in the neck) affects function in both arms, not just the symptomatic side. The investigators will evaluate 42 patients with different cervical nerve root involvement (C4-5, C5-6, or C6-7) and compare them to 16 control subjects with non-specific neck pain. The assessments will measure muscle strength, sensory function, hand performance, pain levels, and psychological factors. These evaluations may contribute to the development of rehabilitation programs for cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Clinical diagnosis of unilateral cervical radiculopathy at C4-5, C5-6, or C6-7 level
* Diagnosis confirmed by clinical examination and MRI
* Symptoms present for at least 4 weeks prior to enrollment
* Ability to understand and follow study instructions
* Ability to provide informed consent for participation
* For control group: non-specific neck pain without radiculopathy
* Ability to complete required assessments

Exclusion Criteria:

* Systemic disorders
* Neurological disorders (excluding CR)
* Previous spinal surgery
* Acute trauma
* Fracture
* Malignancy
* Osteoporosis
* Rheumatic disease
* Ongoing pharmacological treatment for chronic neck pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study will include patients with cervical radiculopathy (CR) and a control group with mechanical neck pain. Participants aged 18 to 65 years will be recruited from X Hospital. CR diagnosis will be confirmed by medical history, physical examination, and MRI findings. Patients will be categorized into three subgroups based on the affected cervical level: C4-5 (C5), C5-6 (C6), and C6-7 (C7). Exclusion criteria will include systemic or neurological disorders (excluding CR), previous spinal surgery, acute trauma, fracture, malignancy, osteoporosis, rheumatic disease, or ongoing treatment for chronic neck pain. Only patients with neck pain for at least three months will be eligible. MRI findings, dermatome mapping, and physical examination will be used to determine the primary affected level in cases of overlapping symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Single assessment at study enrollment
  Upper extremity muscle strength will be measured using a calibrated digital dynamometer. Measurements will be performed for shoulder flexors, extensors, and abductors, elbow flexors and extensors, wrist flexors and extensors, and forearm supination and pronation. Three consecutive measurements will be taken during maximal isometric contraction for each muscle group while the patient is seated in a standardized position, and the highest value will be recorded in Newtons (N). A 30-second rest period will be provided between measurements. Testing will be conducted bilaterally, with the unaffected side tested first.

SECONDARY OUTCOMES:
Light Touch Sensation | Single assessment at study enrollment
  Light touch sensation will be assessed bilaterally using the Semmes-Weinstein monofilament test kit (North Coast Medical Inc., Gilroy, CA, USA). Testing will follow standardized protocols, starting with the 2.83 filament applied to three specific locations on each hand: thumb, index finger, and little finger. Each monofilament will be applied at a 90-degree angle with sufficient pressure to bend it for 1-1.5 seconds, and repeated three times at each location. Participants will respond "yes" when they feel the stimulus. A threshold will be considered achieved when the patient correctly identifies at least seven out of ten applications. Results will be classified as normal (1.65-2.83), diminished light touch (3.22-3.61), diminished protective sensation (3.84-4.31), loss of protective sensation (4.56-6.65), and unmeasurable sensation (above 6.65). Comparison between affected and unaffected sides will be documented.
Vibration Sense | Single assessment at study enrollment
  Vibration sense will be evaluated using a 128 Hz tuning fork applied to the radial and ulnar styloid processes. Participants will be seated with forearms supported and wrists in neutral position. The tuning fork will be struck and applied to each styloid process, with participants indicating when vibration starts and stops. Three measurements will be taken at each site with 30-second intervals between tests. The duration of perceived vibration will be recorded and averaged. Results will be classified as normal, diminished, or absent based on age-normalized values. Comparison between affected and unaffected sides will be documented.
Upper Extremity Function | Single assessment at study enrollment
  Upper extremity functional level will be assessed using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, a standardized 30-item self-report measure validated for upper extremity symptoms and activity limitations. Each item is scored from 1 (no disability) to 5 (most severe disability), with total scores converted to a 0-100 scale. Higher scores indicate greater disability. The questionnaire will be completed by participants at the study enrollment visit.RetryClaude can make mistakes. Please double-check responses.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Beykent University, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No